CLINICAL TRIAL: NCT00024271
Title: Phase II Trial Of Combined Resection, Intraperitoneal Chemotherapy, And Whole Abdominal Radiation For Treatment Of Peritoneal Mesothelioma
Brief Title: Surgery, Chemotherapy, and Radiation Therapy in Treating Patients With Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068907; CPMC-IRB-13799; NCI-G01-2015
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2004-01

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Interferon-gamma; Cisplatin; Doxorubicin; Gemcitabine; Mitomycin; Diathermy; Radiotherapy

INTERVENTIONS:
Biological: recombinant interferon gamma
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: mitomycin C
Procedure: conventional surgery
Procedure: hyperthermia treatment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs directly into the tumor after surgery and combining them with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining surgery, chemotherapy, and radiation therapy in treating patients who have peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, duration of response, and duration of survival of patients with peritoneal mesothelioma treated with surgery, intraperitoneal chemotherapy, and whole abdominal radiotherapy.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients undergo initial surgery, including total omentectomy and excision of gross disease. Approximately 3-4 weeks after surgery, patients receive intraperitoneal (IP) chemotherapy consisting of doxorubicin IP over 2 hours once weekly on weeks 1, 4, 7, and 10 and cisplatin IP and gemcitabine IP once weekly on weeks 2, 5, 8, and 11. Patients also receive interferon gamma IP once weekly on weeks 13-16.

At approximately week 18-20, patients undergo second-look surgery. Patients with no gross disease receive hyperthermia mitomycin IP and cisplatin IP over 90 minutes.

Approximately 2-4 weeks after second-look surgery, patients undergo radiotherapy 5 days a week for 5-7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant mesothelioma
* Measurable or evaluable disease
* Ineligible for other high-priority study
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* SWOG 0-2
* Karnofsky 60-100%

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 times normal

Renal:

* Creatinine clearance at least 45 mL/min
* BUN less than 1.5 times normal
* No significant calcium abnormalities

Cardiovascular:

* No symptomatic cardiovascular disease
* No New York Heart Association class II, III, or IV heart disease
* No congestive heart failure
* No angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension

Other:

* No significant phosphate, electrolyte, or other metabolic abnormalities (e.g., metabolic acidosis)
* No uncontrolled psychiatric disorder or neurologic disease
* No seizure disorder
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or skin cancer
* No other serious medical or psychiatric illness
* No uncontrolled serious infection
* No senility or emotional instability
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 2 prior chemotherapy regimens
* No more than 1 prior intraperitoneal chemotherapy regimen
* More than 6 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except for nondisease-related conditions (e.g., insulin for diabetes)
* Concurrent steroids for antiemesis, premedication, adrenal failure, or septic shock allowed

Radiotherapy:

* No prior abdominal, pelvic, or lower chest radiotherapy

Surgery:

* Prior surgical resection preceding disease recurrence allowed
* More than 1 week since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Taub, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States